CLINICAL TRIAL: NCT04403529
Title: Evaluating the Clinical Value of Traditional Chinese Medicine in the Adjuvant Therapy of Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Head of Breast Surgery Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZY(2018-2020)-CCCX-2005-04
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: adjuvant therapy; traditional chinese medicine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine (Experimental): 60 days of oral Traditional Chinese Medicine ("prescription for breast cancer" Traditional Chinese Medicine formulation)
  Interventions: Drug: Traditional Chinese Medicine Formulation
- Placebo (Placebo Comparator): 60 days of oral placebo (placebo contains 5% "prescription for breast cancer" Traditional Chinese Medicine formulation and 95% filler)
  Interventions: Drug: Placebo Formulation

INTERVENTIONS:
Drug: Traditional Chinese Medicine Formulation — The "prescription for breast cancer" Traditional Chinese Medicine formulation is a combination of 12 herbal components and it is available in granules form to be dissolved in hot water for consumption.
  Other Names: "prescription for breast cancer" Traditional Chinese Medicine formulation
  Arms: Traditional Chinese Medicine
Drug: Placebo Formulation — Placebo granules contains 5% "prescription for breast cancer" Traditional Chinese Medicine formulation and 95% filler, it is available in granules form to be dissolved in hot water for consumption.
  Other Names: Placebo granules contains 5% "prescription for breast cancer" Traditional Chinese Medicine formulation and 95% filler
  Arms: Placebo

SUMMARY:
This is a prospective, single site, randomized, double-blind Phase III clinical trial to evaluate the clinical value of Traditional Chinese Medicine in the adjuvant therapy of triple-negative breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-70 years old;
* Pathologically confirmed stage I-III breast cancer after early breast cancer surgery, and is confirmed by histopathology to be triple negative breast cancer (estrogen receptor (ER)-negative/ progesterone receptor (PR)-negative/ human epidermal growth factor receptor 2 (HER2)-negative). HER2-negative is defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization test is required by local laboratory testing;
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; life expectancy is ≥ 6 months;
* Has adequate organ function meeting the following criteria: (1) adequate bone marrow function: hemoglobin ≥ 90 g/L (no blood transfusion within 14 days); absolute neutrophil count ≥ 1.5 x 109 /L; platelet count ≥ 100 * 109 /L; (2)adequate liver and kidney function: Alanine Aminotransferase (ALT) ≤ 3×upper limit of normal (ULN), Aspartate Aminotransferase (AST) ≤ 3×ULN, Total Bilirubin (TBIL)≤ 1.5×ULN, serum creatinine ≤ 1×ULN，and with endogenous creatinine clearance rate of >50 ml/min (Cockcroft-Gault formula).
* Participant has completed the last of their post surgical radiotherapy and chemotherapy within the last 6 months before date of enrollment, and no tumor recurrence or metastasis at the time of enrollment.
* Participants voluntarily joined the study, has signed informed consent before any trial related activities are conducted, has good compliance and has agreed to follow-up.

Exclusion Criteria:

* Has bilateral breast cancer;
* Has previous history of additional malignancy, with the exception of adequately treated basal cell carcinoma and cervical carcinoma in situ.
* Has metastatic (Stage 4) breast cancer;
* Has any >T4 lesion (UICC1987) (with skin involvement, mass adhesion and fixation, and inflammatory breast cancer);
* Is pregnant, is breast feeding women, or women of childbearing age who cannot practice effective contraceptives;
* Patients participating in other drug related clinical trials at the same time;
* Has severe organ dysfunction (cardiopulmonary liver and kidney) insufficiency, left ventricular ejection fraction (LVEF) < 50% (cardiac ultrasound); severe cardio cerebral vascular disease within the 6 months previous of randomization (such as unstable angina, chronic heart failure, uncontrolled hypertension with blood pressure>150/90mmgh, myocardial infarction, or cerebral blood vessel); diabetic patients with poor blood glucose control; patients with severe hypertension;
* Has known allergy to study medication;
* Has severe or uncontrolled infection;
* Has a history of psychotropic substance abuse and were unable to abandon drug habits, or those with history of mental disorders;
* The researchers judged patients to be unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years
Difference in quality of life scores as assessed by EORTC QLQ-C30 | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
  Difference in quality of life scores as assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). Higher scores mean a better outcome. An higher scores after treatment compared to baseline mean a better outcome or improvement.
Difference in quality of life scores as assessed by EORTC QLQ-BR23 | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
  Difference in quality of life scores as assessed by European Organisation for Research and Treatment of Cancer quality of life questionnaire-breast cancer module 23 (QLQ-BR23). Higher scores mean a better outcome. An higher scores after treatment compared to baseline mean a better outcome or improvement.

SECONDARY OUTCOMES:
Local recurrence rate | 1,2,3 years
Distant metastasis rate | 1,2,3 years
Overall survival | 3 years
Difference in Syndrome of Traditional Chinese Medicine Evaluation of Traditional Chinese Medicine syndromes | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
Difference in physical fitness evaluation by Eastern Cooperative Oncology Group (ECOG) score | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
  Difference in physical fitness evaluation by Eastern Cooperative Oncology Group (ECOG) score, the score runs from 0 to 5, with 0 denoting perfect health and 5 death.
Difference in physical fitness evaluation by Karnofsky performance score (KPS) | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
  Difference in physical fitness evaluation by Karnofsky performance score (KPS), the score runs from 0 to 100, with 100 denoting perfect health and 0 death.
Adverse events | 2 months from baseline, and follow-up every 3 months afterwards until up to 3 years.
  Incidence and Severity of adverse events according to the Common Terminology Criteria for Adverse Events Version 4.0（CTCAE V4.0）

CONTACTS AND LOCATIONS:
Overall Officials: ZhiMin Shao, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality, China